CLINICAL TRIAL: NCT06110195
Title: A Phase I Study of Xevinapant With Radiation and Concurrent Carboplatin and Paclitaxel in Patients Ineligible for Cisplatin With Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Xevinapant With Radiation and Chemotherapy for Patients With Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0294
Record Dates: First submitted 2023-10-20; First posted 2023-10-31 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Escalation Group Dose Level -1 (Experimental): Participants assigned to this cohort will receive xevinapant 50 mg for 2 out of every 3 weeks (Daily on days 1-14 of a 21-day cycle). They will also receive carboplatin and paclitaxel weekly for 7 doses with radiation (chemoRT).
  An additional 3 cycles of xevinapant will be given after completion of chemoRT.
  Interventions: Drug: Xevinapant; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy
- Escalation Group Dose Level 0 (Experimental): Participants assigned to this cohort will receive xevinapant 100 mg for 2 out of every 3 weeks (Daily on days 1-14 of a 21-day cycle). They will also receive carboplatin and paclitaxel weekly for 7 doses with radiation (chemoRT).
  An additional 3 cycles of xevinapant will be given after completion of chemoRT.
  Interventions: Drug: Xevinapant; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy
- Escalation Group Dose Level 1 (Experimental): Participants assigned to this cohort will receive xevinapant 150 mg for 2 out of every 3 weeks (Daily on days 1-14 of a 21-day cycle). They will also receive carboplatin and paclitaxel weekly for 7 doses with radiation (chemoRT).
  An additional 3 cycles of xevinapant will be given after completion of chemoRT.
  Interventions: Drug: Xevinapant; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy
- Escalation Group Dose Level 2 (Experimental): Participants assigned to this cohort will receive xevinapant 200 mg for 2 out of every 3 weeks (Daily on days 1-14 of a 21-day cycle). They will also receive carboplatin and paclitaxel weekly for 7 doses with radiation (chemoRT).
  An additional 3 cycles of xevinapant will be given after completion of chemoRT.
  Interventions: Drug: Xevinapant; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy
- Dose Expansion (Experimental): Participants assigned to this cohort will receive xevinapant at the dose found during escalation phase of study for 2 out of every 3 weeks (Daily on days 1-14 of a 21-day cycle). They will also receive carboplatin and paclitaxel weekly for 7 doses with radiation (chemoRT).
  An additional 3 cycles of xevinapant will be given after completion of chemoRT.
  Interventions: Drug: Xevinapant; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Xevinapant — Given orally during study treatment on days 1-14 of a 21-day treatment cycles. It will be given continuously during treatment with carboplatin, paclitaxel, and radiation (chemoRT). After completely of the chemoRT dosing, an additional 3 cycles of Xevinapant along will be given.
Drug: Carboplatin — Given with radiation weekly for 7 doses.
Drug: Paclitaxel — Given with radiation weekly for 7 doses.
Radiation: Radiation Therapy — Radiation will be given together with paclitaxel and carboplatin for 7 weeks.

SUMMARY:
The goal of this clinical trial is to determine the best safe dose of xevinapant that can be given in combination with chemotherapy and radiation in patients with head and neck cancer. Up to 4 doses of xevinapant will be tested in the dose escalation portion of the study. After the best safe dose is found during escalation, an additional group of participants will be enrolled at that dose to learn more about the treatment combination (dose expansion).

The main question[s] it aims to answer are:

* what is the maximum safe dose that can be given
* what dose should be used in subsequent (phase 2) trials

Participants will receive xevinapant in combination with paclitaxel and carboplatin chemotherapy and radiation. Treatment will be given in 3-week cycles for 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of squamous cell carcinoma of the head and neck (HNSCC) of the oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, or sinuses.

   * Patients with oropharynx cancer need p16 determination by immunohistochemistry (where positive is defined as greater than 70% strong nuclear or nuclear and cytoplasmic staining of tumor cells).
   * Oral cavity, larynx, hypopharynx, or p16-negative oropharynx cancer must be stages T1-2N1-3 or T3-4N0-3 (AJCC 8th edition). Sinus primary must be T4bN0-3 not amenable to surgical resection.
   * P16-positive oropharynx cancer patients, stages T1-2N1-3 or T3-4N0-3 (AJCC 8th edition staging).
2. The patient has unresected, measurable disease as defined by the presence of at least one measurable lesion per RECIST 1.1.
3. Age >= 18 years of age
4. Patients must have a contraindication to cisplatin
5. Performance Status of 0-2
6. Adequate hematologic function

   * White Blood Cell Count (WBC) >= 2000 cells/mm3
   * Absolute neutrophil count (ANC) >= 1,500 cells/mm3
   * Platelets >= 100,000 cells/mm3
   * Hemoglobin >= 9.0 g/dL
7. Adequate renal function was defined as follows: Creatinine clearance (CrCl) > 30 mL/min
8. Adequate hepatic function

   * Total bilirubin <= 1.5 x upper limit of normal (ULN) (except patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL)
   * aspartate aminotransferase (AST) and alanine transaminase (ALT) <= 2.5 x upper limit of normal (ULN)
9. For women of childbearing potential (e.g. uterus present and menstruating), a negative serum pregnancy test within 14 days prior to registration.
10. Willingness to agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of joining the study until 6 months after completing chemotherapy treatment or 3 months after last dose of xevinapant, whichever is the latest.
11. Patients with a history of hepatitis B or C infection are eligible if they have an undetectable viral load.
12. Ability to understand and the willingness to sign a written informed consent document.
13. Availability of tumor tissue for research analysis. Patients who do not have adequate tissue available will need to undergo a new biopsy prior to enrollment on study.

Exclusion Criteria:

1. Definitive clinical or radiologic evidence of distant (beyond cervical lymph node and neck tissue) metastatic disease.
2. Carcinoma of the neck of unknown primary site of origin
3. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable if not within < 3 years
4. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
5. Severe, active co-morbidity defined as follows:

   * History of bone marrow transplant and organ transplant, including allogeneic stem cell transplantation.
   * Unstable angina requiring hospitalization in the last 6 months.
   * New York Heart Association Functional Classification III/IV.
   * Myocardial infarction within the last 6 months.
   * Persistent Grade 3-4 electrolyte abnormalities that cannot be reversed despite as indicated by repeat testing.
   * Ongoing active infection associated with symptoms and/or requires antibiotic therapy at the time of initiation of treatment.
6. Pregnancy and nursing females, if applicable.
7. Receipt of live vaccinations within 28 days prior to study start.
8. Patients who are receiving any other investigational agents.
9. Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to xevinapant, carboplatin, or paclitaxel.
11. Patients taking prohibited medications and those requiring close monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Determine best safe dose of xevinapant when given in combination with radiation and chemotherapy | 21 days

SECONDARY OUTCOMES:
Progression Free Survival | 5 years
  Time from registration to the date of first documented disease progression based on RECIST v1.1, clinical progression, or death due to any cause, whichever occurs first.
Number of side effects seen when xevinapant is given in combination with radiation and chemotherapy | 21 days
Overall Survival | 5 years
  Time between the date of registration and the date of death.
Locoregional failure | 5 years
  Time from registration to the date of first documented disease progression based on RECIST v1.1 in the head and neck.
Distant Failure | 5 years
  Time from registration to the date of first documented disease progression based on RECIST v1.1 below the clavicles.
Response Rate | 5 years
  Complete or partial response per RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ari Rosenberg, ND, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States